CLINICAL TRIAL: NCT05788601
Title: Dapiglutide for the Treatment of Obesity (DREAM): a Randomised, Double-blind, Placebo-controlled, Investigator-initiated Trial
Brief Title: Dapiglutide for the Treatment of Obesity
Acronym: DREAM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Zealand Pharma (Industry)
Responsible Party: Principal Investigator, Filip Krag Knop, Principal Investigator, Clinical Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The 'DREAM' trial; 2022-501649-54-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-02-07; First posted 2023-03-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Inflammation
Keywords: Gut barrier function
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Intervention Model Description: Three arms: 12 weeks of 4 mg and 6 mg dapiglutide and placebo
Who Masked: Participant, Investigator
Masking Description: To ensure blinding, the placebo arm is split between 4 mg and 6 mg placebo, making the randomisation sequence 2:2:1:1 (e.i. 2x 4 mg dapiglutide, 2x 6 mg dapiglutide, 1x 4 mg placebo and 1x 6 mg placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (4 mg and 6 mg) (Placebo Comparator): Abdominal s.c. self-administration of placebo content once weekly for 12 weeks. To ensure double-blinding, the placebo arm is divided into a 4-mg and 6-mg arm. But both placebo arms are pooled during data analysis.
  Interventions: Drug: Placebo
- 4 mg dapiglutide (Active Comparator): Abdominal s.c. self-administration of 4 mg dapiglutide once weekly initiated at 2 mg and up-titrated after three weeks until the remaining nine weeks of treatment (12 weeks in total)
  Interventions: Drug: Dapiglutide
- 6 mg dapiglutide (Active Comparator): Abdominal s.c. self-administration of 6 mg dapiglutide once weekly initiated at 2 mg and up-titrated after three weeks to 4 mg and again to 6 mg after six weeks until the remaining six weeks of treatment (12 weeks in total)
  Interventions: Drug: Dapiglutide

INTERVENTIONS:
Drug: Dapiglutide — GLP-1/GLP-2 receptor agonism
  Other Names: ZP7570
  Arms: 4 mg dapiglutide; 6 mg dapiglutide
Drug: Placebo — Placebo
  Arms: Placebo (4 mg and 6 mg)

SUMMARY:
This study is an investigator-initiated, proof-of-concept, randomised, double-blind, placebo-controlled, parallel-group, single-centre clinical trial investigating the body weight loss potential of dapiglutide, a dual GLP-1R/GLP-2R agonist, administered subcutaneously once weekly. The study will investigate the efficacy of once-weekly subcutaneously administered of 4 mg and 6 mg dapiglutide versus placebo in 54 obese individuals (BMI >30 kg/m2) during a 12-week treatment period.

DETAILED DESCRIPTION:
In total, 54 obese participants with a body mass index (BMI) of ≥ 30 kg/m² are randomised to either treatment with the investigational medicinal product (IMP), being either dapiglutide 4 mg, dapiglutide 6 mg, or placebo for 12 weeks. To ensure blinding, the placebo arm is split between 4 mg and 6 mg placebo, making the randomisation sequence 2:2:1:1. The trial encompasses a 3-week screening period containing a screening visit (V1) to assess eligibility, followed by a randomisation visit (V2) and subsequently a 12-week treatment period concluded with a 4-week follow-up period. The IMP is subcutaneously administered in the abdomen once weekly from week 0 (V2) until week 12 (V14). The IMP is initiated at 2 mg once-weekly and up-titrated every third week with 2 mg until the respective trial doses are reached in each arm. Hereafter, the participants are kept at the dose level for the remainder of the trial (from week 3 and week 6 for the 4 mg and 6 mg doses, respectively). To reduce dropout in cases of low tolerability of the IMP, the investigator can postpone up-titration or down-titrate if judged necessary for participant retention or safety. The trial schedule will consist of five on-site visits, including screening, randomisation and a safety follow-up visit (four weeks after end of treatment (EOT)), in addition to a minimum of 10 telephone consultations. Therefore, the maximum trial duration is 16 weeks. For exploratory purposes, participants are invited to participate in a gastroduodenoscopy sub-study obtaining gastric and duodenal biopsies before and after treatment with IMP. A maximum of 7 participants from each treatment arm (total n=21) participate in this sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* BMI ≥ 30 kg/m²
* History of at least one attempt to lose body weight

Exclusion Criteria:

* A self-reported change in body weight ≥ 5% within the last 90 days prior to the screening visit
* Treatment with any therapy, including endoscopic procedures and/or medication (e.g. liraglutide, bupropion/naltrexone and orlistat), intended for weight management within 90 days prior to screening
* Previous, current, or planned (during the trial period) obesity treatment with surgery or a weight loss device < 1 year prior to screening
* Glycated haemoglobin (HbA1c) ≥ 48 mmol/mol
* History of type 1 diabetes or type 2 diabetes
* Treatment with glucose-lowering agents within 90 days prior to screening
* Compromised kidney function (estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2) at screening
* Known liver disease (except for non-alcoholic fatty liver disease) and/or elevated plasma alanine aminotransferase (ALT) > three times the upper limit of normal at screening
* History of acute and/or chronic pancreatitis
* History and/or family history of medullary carcinoma and/or multiple endocrine neoplasia syndrome
* Inflammatory bowel disease
* Any history of colon cancer or intestinal polyps
* Any history of intestinal stenosis
* History of any other cancers (except margin-free resected cutaneous basal or squamous cell carcinoma or adequately treated in situ cervical cancer) unless disease-free state for at least five years
* Uncontrolled thyroid disease as per discretion of the investigators
* Any of the following: myocardial infarction, stroke, hospitalisation for angina and transient ischaemic attack within the last 60 days prior to screening
* Class IV heart failure according to the New York Heart Association
* Any concomitant disease or treatment that, at the discretion of the investigators, might jeopardise the participant's safety during the trial
* Alcohol/drug abuse as per discretion of the investigators
* Known or suspected hypersensitivity to the trial product or related products
* Previous treatment with the trial product
* Administration of an investigational drug within 90 days prior to screening
* Simultaneous participation in any other clinical intervention trial
* Mental incapacity or language barriers that preclude adequate understanding or cooperation, or unwillingness to comply with trial requirements
* Use of GLP-1RA, GLP-2RA, dipeptidyl peptidase 4 (DPP) inhibitors, human growth hormone, somatostatin, or analogues thereof, within three months prior to screening
* Known radiation enteritis or significant villous atrophy, e.g., due to active coeliac disease or inflammatory bowel disease
* Regarding fertile men and women:

  * Women who are pregnant, breastfeeding, intend to become pregnant or are of childbearing potential will not be included in the study
  * Sterilised or postmenopausal women (> 12 months amenorrhoea or females ≥ 60 years of age) can be included
  * The following contraceptive methods are considered adequate for study enrolment of male participants: Surgically sterilised or willing to refrain from sexual intercourse from screening and until completion of the follow-up visit, or, if sexually active, condom usage and partner-practised contraception during the trial, i.e., from screening to the last visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight (kg) | From week 0 (baseline) to week 12 (end of treatment)
  %-point

SECONDARY OUTCOMES:
Body weight reduction ≥ 5% | From week 0 (baseline) to week 12 (end of treatment)
  count (yes/no)
Body weight reduction ≥ 10% | From week 0 (baseline) to week 12 (end of treatment)
  count (yes/no)
Change in fasting serum/plasma concentrations of gut permeability biomarker (LPS-binding protein (LBP)) | From week 0 (baseline) to week 12 (end of treatment)
  %-point
Change in fasting serum/plasma concentrations of inflammation markers (hs-CRP and IL-6) | From week 0 (baseline) to week 12 (end of treatment)
  %-point

OTHER OUTCOMES:
Body weight reduction ≥ 15% | From week 0 (baseline) to week 12 (end of treatment)
  count (yes/no)
Change in BMI (kg/m2) | From week 0 (baseline) to week 12 (end of treatment)
  %-point
Change in systolic blood pressure (mmHg) | From week 0 (baseline) to week 12 (end of treatment)
  %-point
Change in diastolic blood pressure (mmHg) | From week 0 (baseline) to week 12 (end of treatment)
  %-point
Change in resting heart rate (beats per minute) | From week 0 (baseline) to week 12 (end of treatment)
  %-point
Change in body composition as measured by bioimpedance | From week 0 (baseline) to week 12 (end of treatment)
  %-point
Change in FibroScan®-assessed liver steatosis (dB/m) | From week 0 (baseline) to week 12 (end of treatment)
  %-point
Change in FibroScan®-assessed liver fibrosis (kPa) | From week 0 (baseline) to week 12 (end of treatment)
  %-point
Change in Fatty liver index score (FLI) | From week 0 (baseline) to week 12 (end of treatment)
  %-point (FLI score: Range interval 0-100, < 30 negative likelihood of fatty liver and >60 positive likelihood of fatty liver)
Change in fibrosis 4 score (FIB-4) | From week 0 (baseline) to week 12 (end of treatment)
  %-point (score of <1.30 = low risk; 1.30-2.67 = intermediate risk; >2.67 = high risk of advanced fibrosis)
Change in the 36-Item Short Form Survey | From week 0 (baseline) to week 12 (end of treatment)
  Score points
Change in IWQOL-Lite-CT | From week 0 (baseline) to week 12 (end of treatment)
  Score points
Number of treatment-emergent AEs | From signed consent form (week -3) to follow-up visit (week 16)
  Counts of events
Number of serious AEs (SAEs) | From signed consent form (week -3) to follow-up visit (week 16)
  Counts of events

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research at Gentofte Hospital
Locations (1):
- Center for Clinical Metabolic Research, Herlev-Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No
At this moment we do not plan to share individual participant data

DOCUMENTS (1):
  • Study Protocol (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT05788601/Prot_000.pdf